CLINICAL TRIAL: NCT02413528
Title: Pilot Study of a Mobile Intervention to Increase Adherence to Asthma Medication Among Adolescents
Brief Title: Pilot Study of a Mobile Asthma Adherence Intervention
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Wireless connectivity challenges with device and mobile app
Sponsor: CoheroHealth (Industry)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014_Fall_2014_Sinai
Record Dates: First submitted 2015-04-07; First posted 2015-04-10 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Asthma
Keywords: Patient Compliance; Mobile Applications
MeSH Terms: conditions — Asthma; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care with Medication Monitoring (Sham Comparator): Patients will be given an inhaler sensor to monitor medication use and a sham version of the mobile app that will not include reminders or incentives.
  Intervention: Inhaler sensor
  Interventions: Device: Inhaler sensor
- Medication Monitoring and Mobile App (Experimental): Patients will be given an inhaler sensor to monitor medication use and a mobile phone application that will send them reminders and provide an opportunity to see their own medication use and win incentives for adherence.
  Interventions: Inhaler sensor and mobile application for asthma adherence
  Interventions: Device: Inhaler sensor; Behavioral: Mobile application for asthma adherence

INTERVENTIONS:
Device: Inhaler sensor — Inhaler sensor strap that tracks inhaler use via a pressure sensitive switch.
Behavioral: Mobile application for asthma adherence — Mobile phone application that sends reminders, allows patients to see their medication use, and provides points and other incentives for medication use.
  Arms: Medication Monitoring and Mobile App

SUMMARY:
The purpose of this study is to assess the use of a mobile health intervention to improve adherence to asthma medication among adolescents. The intervention consists of an inhaler sensor strap to monitor asthma inhaler use and a mobile phone application to remind and incentivize patients to use their medication. This study will assess medication use throughout the study in patients who receive a mobile app with reminders and asthma control as measured by the ACT [asthma control test].

ELIGIBILITY:
Inclusion Criteria:

* Age 11-19
* Asthma diagnosis
* Currently on a daily controller HFA (hydrofluoroalkane) medication for Asthma
* English-speaking
* Has a smartphone or access to a smartphone or tablet

Exclusion Criteria:

* Pregnant
* Foster Care
* Emancipated minor

Ages: 11 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Real-time medication adherence in patients receiving reminders and incentives compared to standard care. | 12 weeks
  Analysis of real-time medication use data in the experimental [app + sensor] arm vs the sensor only arm.

SECONDARY OUTCOMES:
Asthma control in patients receiving reminders and incentives compared to standard care (Analysis of the ACT [asthma control test]) | 12 weeks
  Analysis of the ACT [asthma control test] at baseline and follow up for patients in each arm to assess changes in asthma control with use of the mobile app.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Ting, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Michael M Parides, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai

IPD SHARING:
Plan to Share IPD: No